CLINICAL TRIAL: NCT00357201
Title: Evaluation of the Efficacy of T1675, a Per Os Omega 3 and Omega 6 Polyunsaturated Essential Fatty Acid Dietary Formulation Versus Placebo in Patients With Bilateral Treated Moderate Dry Eye Syndrome
Brief Title: Efficacy of T1675 Versus Placebo in Patients With Bilateral Treated Moderate Dry Eye Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LT1675-PIICA-04/04 PHASE II
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Last update posted 2006-07-27 (Estimated); Status verified 2006-07

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Dietary Supplements

INTERVENTIONS:
Drug: Food supplement (T1675)

SUMMARY:
To evaluate the efficacy of a 6-month (± 14 days) dietary supplementation period with T1675, a per os omega 3 and omega 6 polyunsaturated essential fatty acid dietary formulation, versus placebo in patients with bilateral treated moderate dry eye syndrome

DETAILED DESCRIPTION:
The aim of the present study is to evaluate the efficacy of a 6-month (± 14 days) dietary supplementation period with T1675 versus placebo in patients with bilateral moderate dry eye syndrome already treated with tear substitutes, and to point out, through several parameters, the best efficacy parameter that could be used for a future clinical phase III study.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent.
* Male or female aged from 18 to 90 years old.
* Known treated bilateral dry eye.
* Dry eye syndrome confirmed by ocular examination with a fluorescein and/or lissamine green staining, BUT and Schirmer, performed within the last 12 months before Inclusion Visit, for both eyes.
* Bilateral symptomatology suggestive of dry eye defined by: at least one of the following ocular symptoms suggestive of dry eye (burning, stinging, dryness feeling, sandy and/or gritty sensation, light sensitivity, reflex tearing, ocular fatigue) and Questioning on patient's feeling (score >=3).
* Fulfilling the following criteria of dry eye syndrome in both eyes defined by: Keratoconjunctivitis defined by a lissamine green score ≥ 4 (Van Bijsterveld score) and Schirmer test <= 10 mm in 5 min or BUT < 10 s

Exclusion Criteria:

* severe dry eye symptom
* eyelid dysfunction
* severe progressive rosacea
* any relevant ocular anomaly interfering with ocular surface
* best corrected far visual acuity <= 1/10
* history of ocular allergy
* traumatism, infection, inflammation within last 3 months
* ocular surgery and laser within the last 3 months
* lasik, laser, PKR within the last 12 months
* contact lenses
* any concomitant nutritive supplementation, vitamins
* any topical concomitant treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-11; Study Completion 2005-05

PRIMARY OUTCOMES:
Total score of the lissamine green staining test in the right eye on Day 168 (Month 6).

SECONDARY OUTCOMES:
Total score of the lissamine green staining test in the right eye on Day 0, Day 28 (Month 1), Day 84 (Month 3), Month 12, Month 18, Month 24, Month 30, and Month 36
Global efficacy
Tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Catherine CREUZOT-GARCHER, Professor, Principal Investigator — CHU of Dijon, France